CLINICAL TRIAL: NCT06679608
Title: Prospective Longitudinal Multicentric Study to Evaluate Syde® Digital Endpoints in Healthy Adults
Acronym: Syde-CAR
Status: Active, not recruiting | Type: Observational
Sponsor: SYSNAV (Industry)
Responsible Party: Sponsor
Other Study IDs: PR5030-72; 2024-A01925-42 (Other: ANSM)
Record Dates: First submitted 2024-10-25; First posted 2024-11-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to constitute a longitudinal Syde® digital health technology (DHT) dataset to serve as a healthy adult reference for Syde® digital variables development and validation. Subjects will be assessed every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 65 years old
* Signed informed consent
* Subjects with a reported BMI ≥ 17 and ≤ 35
* Subject with unlimited internet connection at home and authorizing automatic data upload
* Subject willing and able to comply with all study procedures including:

  * baseline data and questionnaires data entry on EDC (electronic data capture) throughout the study
  * Syde® related procedures
* Subject confirming to be affiliated to, or beneficiary from, a social security category

Exclusion Criteria:

* Elite athletes (at a national level)
* Pregnant women
* Presence of an orthopedic, neuromuscular, or neurological pathology affecting walking gait quality or requiring a walking aid
* Subjects reporting to have an incapacity or invalidity or to be affected by a chronic disease which can affect their activity and/or their lower limb function
* Subjects reporting to have undergone recent surgical procedures, trauma (within 6 months), or affected by a disease or condition affecting lower limb function within 3 weeks before their inclusion

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be initially provided with information on the study through Ethics Committee validated advertising supports (paper and electronic posters and flyers). These supports will be displayed and distributed by the investigational sites.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Longitudinal change of SV95C (stride velocity 95th centile) | 2 years
  Change of SV95C between baseline and Month 6, Month 12, Month 18 and Month 24.

SECONDARY OUTCOMES:
Assess the transversal adherence of the Syde® device in healthy adults | Baseline
  * Number of subjects reaching the defined threshold of recording hours during the protocol defined period at baseline
  * Number of days necessary to reach the defined threshold of recording hours at baseline during the protocol defined period at baseline
Assess the transversal acceptability of the Syde® device in healthy adults | Baseline
  Usability score at baseline
Assess the longitudinal adherence of the Syde® device in healthy adults | 2 years
  * Change in number of subjects reaching the defined threshold of recording hours during the protocol defined periods between baseline and Month 6, Month 12, Month 18, Month 24
  * Change in number of days necessary to reach the defined threshold of recording during the protocol defined periods between baseline and Month 6, Month12, Month 18, Month 24
Assess the longitudinal acceptability of the Syde® device in healthy adults | 2 years
  Change in usability score between baseline and Month 24
Assess the reliability of Syde® in healthy adults | 2 years
  Reproducibility assessed by ICC (Intra-Class Correlation) and Bland and Altman analysis at each timepoint
Evaluate in this healthy adult cohort the transversal effect on Syde® digital endpoints of gender | Baseline
  Correlation between Syde® derived endpoints and gender. The Syde® derived endpoints will include the SV95C (stride velocity 95th centile).
Evaluate in this healthy adult cohorts the transversal effect on Syde® digital endpoints of age | Baseline
  Correlation between Syde® derived endpoints and age. The Syde® derived endpoints will include the SV95C (stride velocity 95th centile) .
Evaluate in this healthy adult cohorts the transversal effect on Syde® digital endpoints of BMI | Baseline
  Correlation between Syde® derived endpoints and BMI. The Syde® derived endpoints will include the SV95C (stride velocity 95th centile) .
Investigate the relationship between changes in Syde® derived endpoints and changes in age | Month 6, Month 12, Month 18, Month 24
  Comparison between changes in Syde® derived endpoints and changes in age between baseline and Month 6, Month 12, Month 18 and Month 24.
Investigate the relationship between changes in Syde® derived endpoints and changes in BMI | Month 6, Month 12, Month 18, Month 24
  Comparison between changes in Syde® derived endpoints and changes in BMI between baseline and Month 6, Month 12, Month 18 and Month 24.

CONTACTS AND LOCATIONS:
Overall Officials: Shotaro Tachibana, Principal Investigator — Hospices Civils de Lyon - Hôpital Femme Mère Enfant (HFME)
Locations (4):
- France (4):
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant (HFME), Bron
  - Hôpital NOVO (Nord-Ouest Val d'Oise), Pontoise
  - CHU ROUEN - Hôpital Charles Nicolle, Rouen
  - SYSNAV, Vernon

IPD SHARING:
Plan to Share IPD: Yes